CLINICAL TRIAL: NCT02548403
Title: Use of Simethicone to Improve the Bowel Cleansing Effects of Polyethylene Glycol With Ascorbic Acid for Colonoscopy
Brief Title: Effect of Simethicone on Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, In-Kyung Yoo, fellow, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Korea University Prep1
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer
Keywords: Bowel preparation; Simethicone; Polyethylene glycol with ascorbic acid
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Simethicone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-Asc (Active Comparator): group 1 (PEG-Asc, N=130) received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure
  Interventions: Drug: PEG-Asc; Drug: PEG-Asc with simethicone
- PEG-Asc with simethicone (Active Comparator): group 2 (PEG-Asc with simethicone, N=130) received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure.Two packs (200 mg/10 mL each) of simethicone (400 mg) was mixed with last 500 mL of additional clear fluid.
  Interventions: Drug: PEG-Asc; Drug: PEG-Asc with simethicone

INTERVENTIONS:
Drug: PEG-Asc — received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure
  Other Names: •Coolprep®; TaeJoon Pharmaceuticals, Seoul, Korea
Drug: PEG-Asc with simethicone — received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure. Two packs (200 mg/10 mL each) of simethicone (400 mg) was mixed with last 500 mL of additional clear fluid.
  Other Names: Coolprep with gasocol® ; TaeJoon Pharmaceuticals, Korea

SUMMARY:
Optimal bowel preparation is essential for colonoscopy efficacy and safety. Mucosal visualization during colonoscopy is often limited by residual stool, bubbles, bile, intraluminal fluid, and debris, which increase the risk of missing flat adenomas or other small lesions.Therefore, intestinal preparation is necessary to remove residual materials prior to endoscopy.

A combined agent, low-dose PEG with ascorbic acid (PEG-Asc), is one low-volume solution commonly used in Korea (Coolprep®; TaeJoon Pharmaceuticals, Seoul, Korea). However, practitioners have noted an increased incidence of bubble formation with this preparation method.

To the investigators knowledge, no previous study has assessed colon preparation in patients administered simethicone.

The purpose of this study was to compare the quality of bowel preparation and compliance between PEG-Asc and PEG-Asc with simethicone. The effectiveness of adding simethicone as an antifoaming agent to improve bowel cleansing for colonoscopy was evaluated in terms of bowel preparation scale and bubble score, and the compliance of both patients and endoscopists was also investigated using a questionnaire.

DETAILED DESCRIPTION:
1. Study design: endoscopist-blinded, prospective, randomized controlled trial
2. Subjects

   - A single-center, randomized, observer-blinded study was performed at Korea University Hospital in Anam. Outpatients were prospectively enrolled. Each group of the patients will receive PEG-Asc or PEG-Asc with simethicone before colonoscopy.
3. Sampling design: Consecutive recruitment of consenting patients
4. Variables Predictor

   1. group 1 (PEG-Asc) received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure;
   2. group 2 (PEG-Asc with simethicone) received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure;Two packs (200 mg/10 mL each) of simethicone (400 mg) was mixed with last 500 mL of additional clear fluid.
5. Primary Outcome: Quality of bowel preparation [Boston Bowel Preparation Scale, bubble score]
6. Secondary Outcome: Patients and endoscopists' compliance[Tolerability, palatability of patient, fatigue score of endoscopist]

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients,
* aged between18 and 80 years undergoing elective outpatient colonoscopy were eligible for the study

Exclusion Criteria:

* patients who had chronic kidney disease,
* severe heart failure(New York Heart Association [NYHA] class III or IV)
* uncontrolled hypertension (systolic pressure ≥170 mm Hg, diastolic pressure ≥100 mm Hg)
* severe constipation
* any bowel resection
* significant gastroparesis, or
* suspected bowel obstruction or perforation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
the quality of the bowel preparation using Preparation Scale | 20 minutes
  Preparation Scale
  Preparation Scale

SECONDARY OUTCOMES:
Completeness of the bowel preparation | 10 minutes
  Patient compliance was recorded by checking the completeness of the prescribed preparation methods including bowel cleansing agent solution and recommended clear liquid.
the patient's tolerability[questionnaire] | 30 minutes before the colonoscopy
  Patients were asked with questionnaires about the symptoms associated with the preparation to assess the patients' tolerability before the colonoscopy. Patients were asked whether they experienced any of the following : abdominal fullness, cramping, nausea, vomiting, sleep disturbance, and overall discomfort, and these symptoms were scored on a 5-point scale where 1 = "none", 2 = "mild", 3 = "moderate", 4 = "severe", and 5 = "very severe".
the endoscopist's tolerability[Visual Analog Score for fatigue] | 10 minutes
  Endoscopist fatigue during colonoscopy was scored using a Visual Analog Scale, ranging from 1-10, where 1 and 10 represented "strongly disagree" and "strongly agree", respectively.

CONTACTS AND LOCATIONS:
Overall Officials: In kyung Yoo, MD, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Korea University College of Medicine, Seoul, Republic of Korea
Locations (1):
- In Kyung Yoo, Seoul, Anamdong 5-ga, Seongbuk-gu, South Korea